CLINICAL TRIAL: NCT03795662
Title: Surviving Pneumonia
Status: Recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Lindegaard Madsen, Associated professor, MD, PhD, Nordsjaellands Hospital
Other Study IDs: Surviving Pneumonia
Record Dates: First submitted 2018-11-09; First posted 2019-01-08 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Diabetes; Immune status; Nutritional status; Physical inactivity; Risk factors
MeSH Terms: conditions — Community-Acquired Pneumonia; Diabetes Mellitus; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples Urine samples Fecal samples Airway samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community-acquired pneumonia: Adults over 18 years old admitted with confirmed community-acquired pneumonia.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Obervational

SUMMARY:
The study aims to explore risk factors for poor prognosis among patients admitted with community-acquired pneumonia (CAP). During a 5-year study period, all patients (aged ≥ 18 years) admitted with CAP at North Zealand Hospital will be invited for inclusion. Questionnaires, anthropometric measures, laboratory tests, and biomaterials will be collected at admission, daily during admission, at discharge and at follow-up. The main clinical outcomes of the study consist of deaths and development of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Infiltrate on chest radiograph plus one or more of the following:

  * Fever (temperature, ≥38.0°C)
  * Hypothermia (<35.0°C),
  * New cough with or without sputum production
  * Pleuritic chest pain
  * Dyspnea
  * Altered breath sounds on auscultation.

Exclusion Criteria:

* Patients unable to give informed consent
* Patients unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) admitted with community-acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of death from any causes | From date of admission until the day of death from any causes, up to 24 months
  Assessed through patient files
Number of participants who develop diabetes | Up to 24 months
  Assessed through patient files and the national registers

SECONDARY OUTCOMES:
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Through patient files
Oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6-month
Number of participants who are readmitted | Up to 6 months
  Through patient files

OTHER OUTCOMES:
Facal sample to assess changes in microbiome | Day 1, 1 month and 6 months
Urine samples to assess metabolomics | Day 1, 1 month and 6 months
Physical activity monitoring (measured by the AX3 accelerometers) | During admission (up to 7 days), 14 days from discharge (an average of 5 days)
Self-reported physical activity by scoring of the international physical activity questionnaire (IPAQ) | Day 1
Muscle strength (measured by hand grip test) | Day 1, discharge (an average of 5 days), 1 months and 6 months
Muscle strength (measured by 30-sec chair stand test) | Day 1 and discharge (an average of 5 days)
Functional capacity (measured by 6-minutes walking test) | Day 1 and discharge (an average of 5 days)
Activities of daily living (measured by Barthel100) | Discharge (an average of 5 days)
BMI | Day 1, discharge (an average of 5 days), 1 month and 6 months
  Weight (kilograms) and height (cm) will be combined to report BMI in kg/m^2
Waist circumference (measured in cm) | Day 1, discharge (an average of 5 days), 1 month and 6 months
Body composition analysis (measured by DEXA scans) | Day 1, discharge (an average of 5 days), 1 month and 6 months
Body composition analysis (measured by bioimpedance) | Daily during admission, discharge (an average of 5 days), 1 month and 6 months
Nutritional status (measured by NRS2002) | Day 1
Concentration of p-phosphate (mmol/l), p-sodium (mmol/l), p-carbamide (mmol/l), p-potassium (mmol/l) | Daily during admission, 1 month and 6 months
  Blood sampling
Concentration of pro- and anti-inflammatory cytokines (IL-6, Il-1ra, IL-18, IL-10, TNF-alpha) | Daily during admission, discharge (an average of 5 days), 1 month and 6 months
Immune cell phenotyping to identify cell counts various T-cells, B-cells, NK-cells and monocytes | Day 1 and discharge (an average of 5 days)
  Flow cytometry on whole blood
Concentration of blood lipids | Day 1, discharge (an average of 5 days), 1 month and 6 months
  Blood sampling
Scoring of the Charlson Comorbidity Index to predict 10-year survival | Day 1
  Scale ranges from 0 to 33 points to predict survival (%)
Oral status (determined by revised oral assessment guide) | Day 1
Dysphagia screening (eating assessment tool 10) | Day 1
Quality of life (EQ-5D-5L) | Day 1, discharge (an average of 5 days), 1 month and 6 months
Glycemic control during oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
Glucagon concentration during oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
  Blood sampling
Insulin concentration during oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
  Blood sampling
C-peptide concentration during oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
  Blood sampling
GLP-1 concentration during oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
  Blood sampling
GLP-2 concentration during oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
  Blood sampling
GIP concentration during oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
  Blood sampling
Insulin sensitivity index (Matsuda) based on oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
Insulin secretion index based on oral glucose tolerance test | Day 1, discharge (an average of 5 days), 1 month and 6 months
Concentration of galectin-3 (ng/ml), sST2 (ng/ml), and troponins (ng/ml) | Daily during admission, 1 month and 6 months
  Blood sampling
Concentration of NT-proBNP (ng/l) | Daily during admission, 1 month and 6 months
  Blood sampling
Z-value of left ventricle (LV) out of echocardiography | Discharge (an average of 5 days), 1 month and 6 months
  Z-value LV
Z-value of right ventricle (RV) out of echocardiography | Discharge (an average of 5 days), 1 month and 6 months
  Z-value RV
Z-value of left atrium (LA) out of echocardiography | Discharge (an average of 5 days), 1 month and 6 months
  Z-value LA
Shortening fraction (SF) measured in echocardiography | Discharge (an average of 5 days), 1 month and 6 months
  SF (%)
Ejection fraction (EF) measured in echocardiography | Discharge (an average of 5 days), 1 month and 6 months
  EF (%)
Valvular insufficiency measured in echocardiography | Discharge (an average of 5 days), 1 month and 6 months
  Aorta valve regurgitation, pulmonary valve regurgitation, tricuspid valve regurgitation and mitral valve regurgitation (no, minimal, moderate, severe)
Heart rate of 12-lead resting ECG | Daily during admission (up to 5 days)
  bpm
Rhythm during 12-lead resting ECG | Daily during admission (up to 5 days)
  Sinus rhythm yes/no
Axis of the QRS complex out of the 12-lead resting ECG | Daily during admission (up to 5 days)
  Degree
Duration of PQ interval out of the 12-lead resting ECG | Daily during admission (up to 5 days)
  ms
Duration of the QRS complex out of the 12-lead resting ECG | Daily during admission (up to 5 days)
  ms
Number of cardiac events | From date of admission up to 24 months
  Assessed through patient files and the national registers
Sputum samples to assess glucose and lactate concentration (measured by ABL) | On admission, 1 month and 6 months
Sputum samples to evaluate drug resistance and O2 content | On admission, 1 month and 6 months
Forced vital capacity (FVC) during spirometry | Discharge (an average of 5 days)
  Litre
Forced expiratory volume in 1 second (FEV1) during spirometry | Discharge (an average of 5 days)
  Litre
FEV1% predicted during spirometry | Discharge (an average of 5 days)
Chest x-ray to image inflammation of the lungs | On admission, 1 month and 6 months
Early Warning Score (EWS) to identify patients at risk of deterioration in hospital | Daily during admission (up to 5 days)
HbA1c to assess the average blood glucose levels 3 months before admission | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Lindegaard, Assoc. Prof, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Department of Pulmonary and Infectious Diseases, Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryrso CK, Hegelund MH, Dungu AM, Faurholt-Jepsen D, Pedersen BK, Ritz C, Krogh-Madsen R, Lindegaard B. Association between Barthel Index, Grip Strength, and Physical Activity Level at Admission and Prognosis in Community-Acquired Pneumonia: A Prospective Cohort Study. J Clin Med. 2022 Oct 27;11(21):6326. doi: 10.3390/jcm11216326. PMID 36362554